CLINICAL TRIAL: NCT00448695
Title: Phase 1 Study of MRI Targeted Focal Laser Thermal Therapy of Biopsy Confirmed Prostate Cancer
Brief Title: MRI Targeted Focal Laser Thermal Therapy of Biopsy Confirmed Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. John Trachtenberg, University Health Network
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRTA06-1
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: MRI; Laser Thermal Therapy; Focal Ablation; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: MRI Targeted Focal Thermal Therapy of Prostate Cancer — The Interstitial Laser Thermal Therapy (LTT) procedure is similar to brachytherapy, with fibers and probes inserted trans-perineal using transrectal ultrasound guidance. Patients will be under general anesthetic, and the procedure is expected to last 3 hours. Patients will be able to return home the day of the procedure.

SUMMARY:
The objective of this study is to establish the safety of MRI targeted laser thermal treatment for men with biopsy confirmed early stage low grade single sector prostate cancer.

DETAILED DESCRIPTION:
This is a single center, single arm, open-label Phase I study to establish the safety of interstitial laser thermal therapy (ILTT) in patients with a single site of low grade (Gleason <7) prostate cancer who have not yet received treatment for their cancer. No control group will be utilized and all patients will receive laser thermal therapy. The patient will undergo multimode MRI to determine if a single site of prostate cancer can be localized by this technique and to localize the tumor in 3 dimensions within the prostate. A multicore (12 + cores) mapping transrectal ultrasound guided biopsy of the prostate would then confirm that no other sites of cancer exist.

Each patient will complete quality of life and performance questionnaires. ILLT will be performed under general anesthetic in a procedure similar to brachytherapy, using transrectal ultrasound to guide insertion of the laser and monitoring probes into the sector containing the cancer as visualized by the MR scan. Following the procedure, patients will be assessed for clinical signs of urinary, rectal, and erectile complications and will complete validated self-assessment tools on these functions. MRI at 7 days and MRI and biopsy at 6 months will be used to assess the extent of tissue effect and presence of cancer due to ILTT. Patients will remain on standard Watchful Waiting surveillance for any further sign of disease progression. ILLT will not restrict any future treatment of prostate cancer.

To minimize the treatment risk, participants in the trial will be staged according to location of the disease in the prostate. The first 3 participants recruited to the trial will have targeted loci well separated from the urethra, erectile nerves and the rectum, and so treatment in this region poses minimal risk of injury to these vital structures. Lesions sizes measured in this initial stage will be used in planning fiber placement in the three remaining stages, in which fiber placement is closer to critical structures such as the urethra (Stage 2), erectile nerves (Stage 3) and rectum (Stage 4).

ELIGIBILITY:
Inclusion Criteria:

* Men > 18 years of age;
* Histologically-proven prostate carcinoma;
* Prostate cancer clinical stage T1c
* Only one sector of the prostate demonstrating prostate cancer with no more than 1 core positive
* Gleason score <7 ;
* Each core must range between of 10 to 50% adenocarcinoma.
* Prostate MRI must confirm area suspicious for cancer in the sector of the positive biopsy;
* A minimum of six (6) weeks between the prostate biopsy and the Inclusion Visit;
* Prostate specific antigen (PSA) level £ 10 ng/mL
* PORPUS, IPSS, and IIEF complete prior to procedure
* Prostate volume < 60 cc as measured by ultra sound;
* Uroflow >12 cc/sec with post void residual < 100 cc.
* Life expectancy of greater than 5 years, based on co-morbidity not related to prostate cancer.

Exclusion Criteria:Patients with any of the following exclusion criteria will be excluded from study participation:

* Patients who are unwilling or unable to give informed consent;
* Patients with foci location in the Apex of the prostate or isolated transition zone cancers
* Patients who have received androgen suppression therapy
* Patients who have received or are receiving chemotherapy for prostate carcinoma;
* Patients previously treated with surgery to the prostate (traditional, endoscopic or minimally invasive including HIFU, TUNA, RITA, microwave, TURP ,cryotherapy or any curative treatment
* Patients whose has undergone radiation therapy for prostate cancer
* Any condition, or history of illness or surgery that, in the opinion of the Investigator , might confound the results of the study or pose additional risks to the patient (e.g. significant cardiovascular conditions or allergies);
* Patients with a history of non compliance with medical therapy and/or medical recommendations;
* Patients who are unwilling or unable to complete the patient self-assessment questionnaires;
* Myocardial infarction, transient ischemic attack or stroke, within 6 months prior to the study, Unstable or uncontrolled angina, uncontrolled heart failure, or serious uncontrolled ventricular arrhythmias
* Chronic or acute prostititis, neuroginic bladder, urinary tract infection, sphincter abnormalities, or any other symptom that prevents normal micturition.
* Patients who have participated in a clinical study and/or received treatment with an investigational treatment and/or product within the past 90 days;
* All medications that cause a decrease clotting, vasoconstriction or platelet aggregation, must be stopped prior to treatment.
* History of Colon Cancer or Colon Surgery preformed
* If the patient is unable to undergo anesthesia
* Patients with contraindication to MRI (i.e. pacemaker, hip prosthesis, severe claustrophobia, brain aneurysm clip, allergy to MRI contrast agent).
* Any condition, or history of illness that, in the opinion of the investigator will confound or increase the patient risk during the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of: urinary, rectal, erectile function | 1 week, 1 month, 3 months, 6 months post procedure
validated self assessment tools of urinary, rectal, erectile function. | 1 month, 3 months, 6 months post procedure

SECONDARY OUTCOMES:
Lesion size measured with 7-day MRI | One week post procedure
6 month prostate biopsy | 6 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: John Trachtenberg, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada